CLINICAL TRIAL: NCT03333083
Title: Phase 3b, Single Arm, Simplification Study With Dual Therapy Including Lamivudine (300 mg QD) Plus Raltegravir (1200 mg QD) in Virologically Suppressed HIV-1 Infected Patients Experiencing Inconvenience, Toxicity, Negative Impact on Co-morbidities or Risk of Drug-drug Interactions With Their Current Regimen. (RALAM-II Study)
Brief Title: Study With Dual Therapy Including Lamivudine (300 mg QD) Plus Raltegravir (1200 mg QD) in Virologically Suppressed HIV-1 Infected Patients Experiencing Inconvenience, Toxicity, Negative Impact on Co-morbidities or Risk of Drug-drug Interactions With Their Current Regimen
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The reason for the premature termination was the failure to reach the required number of participants.
Sponsor: Judit Pich (Other)
Collaborators: Fundacion Clinic per a la Recerca Biomédica (Other)
Responsible Party: Sponsor-Investigator, Judit Pich, Clinical Research Manager, Hospital Clinic of Barcelona
Organization: Hospital Clinic of Barcelona (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RALAM-II; 2017-000985-31 (EudraCT Number)
Record Dates: First submitted 2017-09-29; First posted 2017-11-06 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: HIV Seropositivity; HIV Infections; HIV-1-infection
Keywords: Lamivudine; Raltegravir
MeSH Terms: conditions — HIV Seropositivity; HIV Infections | interventions — Raltegravir Potassium; Lamivudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Raltegravir + Lamivudine (Experimental)
  Interventions: Drug: Raltegravir; Drug: Lamivudine

INTERVENTIONS:
Drug: Raltegravir — Raltegravir (1200 mg once a day)
Drug: Lamivudine — Lamivudine (300 mg once a day)

SUMMARY:
Phase 3b, single arm, simplification study with dual therapy including Lamivudine (300 mg QD) plus Raltegravir (1200 mg QD) in virologically suppressed HIV-1 infected patients experiencing inconvenience, toxicity, negative impact on comorbidities or risk of drug-drug interactions with their current regimen.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients will be males or females at least 18 years of age. Women of childbearing potential must have a negative pregnancy test within 10 days prior to randomization into the study.
* Patients seropositive for HIV-1 using standard diagnostic criteria.
* Patients experiencing inconvenience, toxicity, negative impact on comorbidities or risk of drug-drug interactions with their current regimen
* Patients virologically suppressed during at least 12 months prior to inclusion (viral load <50 copies/mL).
* Patients who have signed informed consent to participate in the study.

Exclusion Criteria:

* Pregnancy, lactation, or planned pregnancy during the study period.
* Previous failure to an integrase inhibitor-containing regimen.
* Previous failure to a Lamivudine or Emtricitabine-containing regimen.
* Resistance mutations to Lamivudine or integrase inhibitor if any resistance test had been previously performed.
* Any disease or history of disease which, in the opinion of the investigator, might confound the results of the study or pose additional risk to patient treatment.
* Chronic hepatitis B.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-05-03 (Actual); Primary Completion 2020-06-25 (Actual); Study Completion 2020-06-25 (Actual)

PRIMARY OUTCOMES:
Therapeutic failure | 48 weeks
  therapeutic failure at week 48, includes virological failure, change in treatment for any reason, consent withdrawal, loss to follow-up or death

SECONDARY OUTCOMES:
Change from baseline in the reason of change of the antiretroviral treatment in those patients the reason of change was inconenience | 48 weeks
  Changes in quality of life calculated by EQ-5D-5L if reason of switch was inconvenience
Change from baseline in the reason of change of the antiretroviral treatment in those patients the reason of change was neurological toxicity | 48 weeks
  Changes on Pittsburgh Sleep Quality Index for neurological toxicity
Change from baseline in the reason of change of the antiretroviral treatment in those patients the reason of change was cardiovascular toxicity or co-morbidity | 48 weeks
  Changes on plasma lipids cholesterol LDL
Change from baseline in the reason of change of the antiretroviral treatment in those patients the reason of change was cardiovascular toxicity or co-morbidity | 48 weeks
  Changes on plasma lipids cholesterol HDL
Change from baseline in the reason of change of the antiretroviral treatment in those patients the reason of change was cardiovascular toxicity or co-morbidity | 48 weeks
  Changes on plasma lipids triglycerides
Change from baseline in the reason of change of the antiretroviral treatment in those patients the reason of change was skeletal toxicity | 48 weeks
  Changes on dual energy x-ray absorptiometry bone density
Change from baseline in the reason of change of the antiretroviral treatment in those patients the reason of change was digestive toxicity | 48 weeks
  Apperance of any adverse event that resolve their digestive toxicity: as diarrhea or digestive discomfort
Change from baseline in the reason of change of the antiretroviral treatment in those patients the reason of change was drug-drug interactions | 48 weeks
  Proportion of drug-drug interaction with antirretroviral treatment
Therapeutic failure | 24 weeks
Virological failure | 24 weeks
  Defined as two consecutive measurements of plasma viral load above 50 copies/ml
Virological failure | 48 weeks
  Defined as two consecutive measurements of plasma viral load above 50 copies/ml
Proportion of patients with viral load below ultrasensitive HIV-1 RNA detection limit (limit of detection 1 copy/mL) | 48 weeks
Changes from baseline in cholesterol total | 24 weeks
Changes from baseline in HDL | 24 weeks
Changes from baseline in triglycerides | 24 weeks
Changes from baseline in insulin resistance (HOMA-IR) | 24 weeks
Changes from baseline in cholesterol LDL | 24 weeks
Changes from baseline in cholesterol LDL | 48 weeks
Changes from baseline in cholesterol total | 48 weeks
Changes from baseline in cholesterol HDL | 48 weeks
Changes from baseline in triglycerides | 48 weeks
Changes from baseline in and insulin resistance (HOMA-IR) | 48 weeks
Changes from baseline in body fat composition | 48 weeks
Changes from baseline in immune activation markers including CD38 | 48 weeks
Changes from baseline in immune activation markers including HLA-DR | 48 weeks
Changes from baseline in biomarkers of inflammation IL-6, | 48 weeks
Changes from baseline in biomarkers of inflammation high sensitivity C-reactive protein | 48 weeks
Changes from baseline in biomarkers of mononuclear activation SD-14 | 48 weeks
Changes from baseline in biomarkers of mononuclear activation SD-163 | 48 weeks
Changes from baseline in sleep quality (Pittsburgh Sleep Quality Index) | 24 weeks
Changes from baseline in sleep quality (Pittsburgh Sleep Quality Index) | 48 weeks
Change from baseline in EQ-5D-5L | 24 weeks
Change from baseline in EQ-5D-5L | 48 weeks
Incidence of adverse events | 48 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínic i Provincial de Barcelona, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No